CLINICAL TRIAL: NCT00867594
Title: A Single Blind, Open-Label Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of Oral Insulin Formulation in Type 1 Subjects
Brief Title: Effectiveness of Oral Insulin in Unstable Type 1 Diabetes Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Oramed Pharmaceutical Inc. (Industry)
Responsible Party: Dr. Roy Eldor, Hadassah Medical Organization, Jerusalem
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0566-08-HMO-CTIL
Record Dates: First submitted 2009-03-22; First posted 2009-03-24 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2008-03

CONDITIONS: Brittle Type I Diabetes Mellitus

INTERVENTIONS:
Drug: ORMD 0801 — 1 capsule ORMD 0801 3 times a day, before each meal

SUMMARY:
The intent of the proposed study is to assess the potential of oral insulin to mitigate diabetic instability and reduce the frequency and severity of hypoglycemic episodes in patients with type 1 diabetes. Restoring hepatic glycogen stores is critical for the normalization of counter-regulation to hypoglycemia in these patients. Oral insulin can provide a means to increase portal insulin levels, shift the ratio of insulin/glucagon in favor of glycogenesis while sparing the patient the risk of hypoglycemia due to peripheral hyperinsulinemia

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus
* Male or female aged 18-50 years inclusive
* Body weight between 50-100kg and BMI between 18 and 30 kg/m2
* Diagnosed 6 or more months ago, unstable diabetes with frequent episodes of hypoglycemia
* No other medical problems

Exclusion Criteria:

* History or presence of clinical significant gastrointestinal pathology or symptoms, liver or kidney disease or any condition that might interfere with the absorption, distribution, metabolism or excretion of the drug
* Positive pregnancy test or lactation
* Lack of family support
* Unwilling or unable to follow the study protocol
* Concurrent medical problems

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of multi-doses of Oramed oral insulin in people with type 1 diabetes | 15 days

SECONDARY OUTCOMES:
To determine if oral insulin is likely to improve glycemic stability assessed by the reduction of the frequency and severity of hypoglycemic episodes in people with unstable type 1 diabetes | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Roy Eldor, Principal Investigator — Hadassah
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel

REFERENCES:
- [Derived] Eldor R, Arbit E, Corcos A, Kidron M. Glucose-reducing effect of the ORMD-0801 oral insulin preparation in patients with uncontrolled type 1 diabetes: a pilot study. PLoS One. 2013 Apr 9;8(4):e59524. doi: 10.1371/journal.pone.0059524. Print 2013. PMID 23593142